CLINICAL TRIAL: NCT03892096
Title: Development of a Cell Free DNA Assay as a Biomarker for Predicting Early Non-response to Therapy in Metastatic Cancer
Status: Completed | Type: Observational
Sponsor: Cadex Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: CADEX-0001
Record Dates: First submitted 2019-03-21; First posted 2019-03-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Non-Small Cell Lung Carcinoma; Metastatic Colorectal Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Up to 30mL of blood via venipuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Lung Cancer, Colorectal Cancer or Breast Cancer: A total of 750 subjects with lung cancer, CRC and breast cancer will be consecutively enrolled. It is expected that 250 subjects will be lung cancer patients, 250 mCRC patients and 250 breast cancer patients.
  Interventions: Diagnostic Test: Blood-based cell-free cfDNA qPCR assay

INTERVENTIONS:
Diagnostic Test: Blood-based cell-free cfDNA qPCR assay — Up to 30mL of blood via venipuncture

SUMMARY:
Accrue samples for the further development and clinical validation of a blood-based cell-free DNA (cfDNA) quantitative real-time polymerase chain reaction (qPCR) assay as a potential biomarker for early non-response to therapy in stage IV non-small cell lung cancer (NSCLC), colorectal cancer (CRC) and breast cancer (BC).

DETAILED DESCRIPTION:
Most anticancer drugs are effective only in subgroups of patients, and our current understanding of tumor biology does not allow us to predict accurately which patient will benefit from a specific therapeutic regimen. The definitive proof of the effectiveness of a therapy is improvement in clinical symptoms and survival. Imaging is generally used to assess therapeutic effects earlier and more objectively. Current response assessment is based primarily on changes in tumor size as measured by CT or other anatomic imaging modalities.

Cadex Genomics has developed an analytically validated cell-free DNA (cfDNA) quantitative real-time polymerase chain reaction (qPCR) assay that utilizes standard qPCR platforms for processing, this test can reliably obtain results from small blood volumes and possesses exceptionally high analytical sensitivity of circulating cfDNA.

The purpose of this study is to accrue samples for the further development and clinical validation of a blood-based cell-free cfDNA qPCR assay as a potential biomarker for early non-response to therapy in stage IV non-small cell lung cancer (NSCLC), colorectal cancer (CRC) and breast cancer (BC).

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

Documented stage IV NSCLC, SCLC, BC or CRC (can be new diagnosis, persistent or recurrent disease):

BC patients who meet the following criteria:

ER+/HER2- and has failed hormone therapy within the last two years, or ER+/HER2+ or, ER-/HER+ or, HER2-/ER-/PR- (TNBC), and Has ≥ 1 measurable non- bone lesion as measured per RECIST or, If bone only disease, has two or more measurable (> 1 cm by RECIST) predominantly lytic bone lesions

Planned initiation of new systemic first- or second-line treatment or subsequent therapies with chemotherapy, immunotherapy, targeted therapy or combination thereof. Or continuation of the current line of therapy after RECIST/iRECIST evaluation which coincides with end of the cycle of therapy and prior to initiation of the next cycle of therapy.

Imaging to determine RECIST and/or iRECIST criteria:

If baseline blood draw is planned prior to first cycle of a line (1st, 2nd, 3rd etc) of therapy, measurable disease with CT or MRI or PET/CT monitoring should be completed within 4 weeks prior to baseline blood draw.

If baseline test is performed at the completion of a cycle of therapy, CT or MRI or PET/CT monitoring should be completed to coincide with end of cycle of therapy and prior to baseline blood draw.

Planned CT or MRI or PET/CT monitoring for treatment response completed within 8-12 weeks of start of treatment.

Willing and able to donate up to 30mL of blood at each blood draw. Willing and able to provide informed consent.

Exclusion Criteria:

Diagnosis of a secondary malignancy that is not in complete remission. Imaging to determine RECIST and/or iRECIST criteria is not planned or available.

CT or MRI or PET/CT monitoring for treatment response is not planned within 8-12 weeks.

Presence of active autoimmune disease which is under active treatment. DVT, PE, sepsis, or has recovered from any other serious illness within the prior 2 weeks of the baseline blood draw. (Note: Patients who have recovered from similar conditions more than 2 weeks prior to the baseline blood draw would be eligible for the study) If initiating a new line of therapy, patient has received any doses of the new block of therapy before the first designated blood draw.

If continuing current line of therapy after CT, MRI or PET/CT monitoring, patient has received subsequent cycle of therapy before the first designated blood draw.

Performance status ECOG ≥3. Evidence of acute renal failure as determined by current clinical guidelines. NSCLC, SCLC or CRC patients beyond 9 months of the initiation of therapy, on 1st line immunotherapy alone, or combination immunotherapy and chemotherapy regimens. (Note: patients on subsequent lines of therapy (2nd,3rd line etc.) would be eligible at any time point including prior to the 9 months vs those patients on 1st line therapy)..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 750 subjects with Lung Cancer, CRC or BC will be enrolled consecutively into each cancer group. It is expected that each group will enroll 250 subjects each. As each group meets its enrollment goals, that group will close to further enrollment.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
DNA Integrity Index as a predictor of progressive disease in a cohort of metastatic patients (250 Lung Cancer (NSCLC, SCLC), 250 CRC and 250 BC patients as compared to standard RECIST/iRECIST criteria. | Six months to accrue patient for initial development
  A total of 750 subjects (250 stage IV Lung Cancer, IV 250 CRC and IV BC) will be enrolled consecutively into the study. Blood specimens will be collected at the initiation of therapy and 12 to 16 days after the initiation of therapy. A course of therapy is defined as chemotherapy, immunotherapy or oral therapy. Standard baseline RECIST or iRECIST will be recorded before the initiation therapy and again at 9-12 weeks. For those patients who are receiving single agent regimen consisting of immunotherapy alone there will be an additional blood draw prior to administration of the second course of therapy. The Integrity Index will be evaluated for predicting early non-response to therapy as compared to standard RECIST/iRECIST results.

CONTACTS AND LOCATIONS:
Overall Officials: Christer Svedman, M.D. Ph.D., Study Director — Cadex Genomics
Locations (12):
- United States (11):
  - CARTI Cancer Center, Little Rock, Arkansas
  - Sutter Health - Palo Alto Medical Foundation, Sunnyvale, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - IACT Health, Columbus, Georgia
  - University Medical Center, New Orleans, Louisiana
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana
  - Nebraska Cancer Center, Omaha, Nebraska
  - National Translational Research Group LLC, Port Jefferson Station, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Advent Health, Hendersonville, North Carolina
  - Greenville Health System - Prisma Health, Greenville, South Carolina
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No